CLINICAL TRIAL: NCT00108446
Title: Characterization of Pain Processing Mechanisms in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLIN-008-02F
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; visceral hypersensitivity; cutaneous hypersensitivity; lidocaine
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Dextromethorphan; Naloxone; Fentanyl; Lidocaine

INTERVENTIONS:
Drug: dextromethorphan
Drug: naloxone
Drug: fentanyl
Drug: lidocaine

SUMMARY:
This study is being done to collect new information on irritable bowel syndrome, a disease that causes abdominal pain that does get better with treatment or keeps coming back ("chronic"). To better understand what causes the irritable bowel syndrome, we are studying drugs used to treat pain, dextromethorphan, naloxone, fentanyl, and lidocaine. We will study the effects these drugs have on experimental pain.

Dextromethorphan is used in non-prescription cough syrups. Naloxone is used for reversing the effects of narcotic pain relievers. Fentanyl is a narcotic used to treat pain and to make a person relaxed (sedated) before anesthesia. The purpose of this study is to see what kinds of pain are affected by these drugs in persons who have irritable bowel syndrome and persons who do not have this problem.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a common gastrointestinal disorder characterized by chronic abdominal pain and altered bowel function (diarrhea and/or constipation) that effects up to 20% of the United States population. Although the pathophysiology of IBS is unknown, visceral hypersensitivity (i.e., decreased pain thresholds in response to gut distension) is a biological marker of the disorder. The mechanisms that lead to visceral hypersensitivity, however, are currently unknown. As a consequence of our current VA-supported studies, our laboratory has acquired evidence that patients with IBS and visceral hypersensitivity also have cutaneous hypersensitivity in response to experimental thermal pain stimuli. These new findings differ from previous investigations that indicated IBS-associated hypersensitivity is limited to the gut. Rather, our data suggest that patients with IBS have alterations in central pain processing mechanisms that may represent the underlying pathophysiological basis for visceral and cutaneous hypersensitivity. Based on our preliminary data, we propose that alterations in spinal processing mechanisms are similar in patients with IBS to those that have been described for patients with other chronic pain disorders. Cutaneous hypersensitivity is also seen in other chronic pain conditions such as fibromyalgia where altered central pain processing mechanisms have been shown to be responsible for maintaining hypersensitivity. In our current proposal, we hypothesize that IBS patients have increased peripheral and central afferent processing of nociceptive cutaneous and visceral stimuli.

Our objectives are as follows:

* Specific Objective #1. To determine if lidocaine applied to the rectum decreases visceral hyperalgesia, as tested by nociceptive rectal distension.
* Specific Objective #2. To determine if lidocaine applied to the rectum decreases cutaneous heat hyperalgesia to test for the presence or absence of central hyperalgesia in IBS patients.
* Specific Objective #3. To determine the relationships between doses of IV lidocaine, serum levels of IV lidocaine, and their anti-hyperalgesic effects, as tested by rectal distension and cutaneous heat stimulation.

Specific Objective #4. To determine the effect of rectal lidocaine on clinical pain and clinical symptoms of IBS.

The proposed studies will test the central hypothesis using well-controlled sensory stimuli designed to separately evaluate central and peripheral mechanisms. The objectives will be accomplished by systematically applying and comparing pharmacological and psychophysical studies to IBS patients and controls. This application is an extension of the principal investigator's current VA Advanced Career Development Award that examines the neurobiology of visceral hypersensitivity in Persian Gulf veterans who returned home with chronic abdominal pain. The proposed Clinical Research Program will study afferent mechanisms of visceral and cutaneous hypersensitivity in veterans with IBS. Our laboratory is uniquely positioned to use our expertise in psychophysical and pharmacologic evaluation of patients with fibromyalgia to study patients with IBS. The results of this current proposal will lead to larger clinical trials with sodium-channel blockers (i.e., lidocaine, mexiletine) as potential therapeutic agents for veterans with IBS.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women age 18 years or older OR healthy controls
* Patients with diarrhea predominant IBS that meet the *Rome II criteria
* The subject must speak English and be able to give informed consent
* All subjects will be tested in the follicular stage of the menstrual cycle as determined by menstrual history and urine testing
* Functional Bowel Disorder Severity Index score of none (0 points) for controls and moderate (37-110 points) for IBS patients
* Normal baseline EKG

Exclusion Criteria:

* Subject is currently participating in another research protocol that could interfere or influence the outcome measures of the present study
* Subject is unable to give informed consent
* A medical condition that would contraindicate the use of lidocaine (i.e., amide allergy) or a previous history of an abnormal EKG
* Subjects with a positive pregnancy test will be excluded because the use of lidocaine is contraindicated in pregnant women
* Subject is currently taking pain medications, NSAIDs, antihistaminics, antidepressants (tricyclic antidepressants [TCA]/selective serotonin reuptake inhibitors [SSRI]), anti-convulsants, migraine medications, and cough suppressants
* Presence of systemic disease: diabetes, thyroid disease, gastrointestinal/liver disease (other than IBS), collagen vascular disease, focal or systemic neurological disease, malignancy, seropositive for HIV, or documented psychiatric disorders
* Presence of any chronic pain condition including fibromyalgia
* Subject drinks > 2 oz. alcohol/day on a regular basis
* Presence of large, palpable hemorrhoids on digital rectal exam that may alter rectal lidocaine adherence to rectal wall
* Abnormal baseline EKG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- Malcom Randall VAMC, Gainesville, Florida, United States